CLINICAL TRIAL: NCT03119415
Title: Enlisting Peer Cooperation and Prosociality in the Service of Substance Use Prevention in Middle School
Acronym: Prosocial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AA024275
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Social Behavior
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Intervention Model Description: This research is a comparison between the Cooperative Learning program and services as usual. Approximately twelve middle schools will be randomized to a waitlist-control condition. The intervention group will receive training in Cooperative Learning immediately and the waitlist-control group will receive training at the end fo the project. Teachers will be given training on the basics of Cooperative Learning and will be supported in their efforts to implement it in their classrooms. No curricular changes will be required. The initial training will last two or three days and will confirm to the professional development calendar of the intervention schools (selected at random). The implementation of Cooperative Learning is expected to be on-going for the full duration of the project (two years).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooperative Learning (Experimental): Teachers in intervention schools are training in cooperative learning (CL).
  Interventions: Behavioral: Cooperative Learning
- Business as Usual (No Intervention): Schools continue with business as usual.

INTERVENTIONS:
Behavioral: Cooperative Learning — CL is an umbrella term that includes peer tutoring, reciprocal teaching, collaborative reading, and other methods in which peers help each other learn in small groups. CL is not prescriptive but rather is a conceptual framework within which teachers design their own small-group activities. Johnson, Johnson, and Holubec's approach to CL combines positive interdependence with individual accountability, a high degree of face-to-face social interaction among youth, and support for the development of cooperative social skills. The Johnsons' approach offers teachers the combination of specific cooperative activities and the conceptual tools to create their own lesson plans using positive interdependence.
  Arms: Cooperative Learning

SUMMARY:
Students' cooperative and prosocial behavior is vital to their social and academic success and to the quality of a school's social environment. This project will evaluate an instructional technique that could benefit students and schools by encouraging higher levels of prosocial behavior among students and promoting social integration and inclusion, particularly for marginalized students. The instructional technique is called "cooperative learning" which involves students working in groups toward shared academic goals. Previous research indicates that cooperative learning promotes social acceptance and increases academic engagement and achievement. However, it has not been evaluated as a technique to reduce student behavioral problems and promote greater school safety. There is strong reason to believe that it will have these benefits, since cooperative learning brings together students from diverse social groups and provides them the opportunity to work together toward shared goals in a positive setting.

DETAILED DESCRIPTION:
A key contributing factor to the initiation and escalation of substance use during early adolescence is affiliation with deviant peers. These affiliations often arise when socially isolated and rejected youth aggregate and reinforce substance use and other deviant activity within the group (i.e., "deviant peer clustering"). Even though the field has developed a number of efficacious prevention programs, few have demonstrated strong effects on deviant peer clustering. Further, on a national level, substance use among adolescents continues to be high, suggesting that a fresh approach to prevention with a renewed focus on the peer context is needed to create a broad, sustainable public health impact.

Existing programs have proven difficult to disseminate with fidelity, often due to their complex design or the significant expenditures required for curricula, materials, and training. To realize broader public health benefits, an approach that integrates scientific knowledge across domains must be applied to develop and test programs that address root causes of youth substance use, are less complex and expensive to implement, are more flexible and adaptable to local conditions, and once established, can spread.

This proposal represents an approach to prevention in which evolutionary theory provides a unifying theoretical framework, which implies that diverse problems are due to social environments that are unfavorable for the expression of prosocial behaviors, instead eliciting a variety of self-oriented or exploitative behaviors. Systematic efforts to reduce multiple problems among youth (e.g., substance use, risky sex, depression, academic failure, etc.) need to look beyond the immediate issues to the social conditions that make the entire range of problems more likely. Programs should focus on modifying key social environments to nurture prosocial behavior and minimize the toxic or stressful conditions that give rise to behavioral problems in youth.

The investigators propose to integrate a few simple, flexible, and powerful prevention strategies that have proven value in establishing a social context conducive to positive peer group development. This project will apply cooperative learning and behavioral kernels to reduce social rejection and isolation, promote new friendships among youth from different social groups, and encourage greater levels of prosocial behavior. This should create a positive feedback loop in which the social and behavioral processes "amplify" one another to bring significant change to the school social context, interrupting deviant peer clustering and addressing a key root cause of escalations in substance use and related problem behavior. With this approach, the investigators anticipate a simple, straightforward implementation, greater sustainability, and opportunities for the program to spread through sharing of best practices among teachers. This project will conduct a small-scale randomized controlled trial involving 12 middle schools in the state of Oregon.

Aim 1a of the project is to evaluate the main effects of the program on both prosocial behavior and substance use. The investigators will also examine effects on secondary outcomes, including delinquent and high-risk sexual behavior, teasing and harassment, depression, school attendance, and academic achievement. The project will include an assessment of program fidelity, which will be incorporated into data analyses. Aim 1b of the project is to explore links among peer rejection, prosocial behavior, and substance use over time in an attempt to determine the direction of effects, which can inform both developmental theory and future intervention design.

Aim 2 will evaluate social network changes as a mediator of intervention effects. The investigators will use longitudinal social network analysis (RSiena) to examine a variety of processes as mediators of effects, including deviant peer clustering. This analyses will provide (1) fresh insight into the processes by which deviant peer groups form, how they impact substance use and related problem behavior, and the ways in which prevention programs may be able to counteract or interrupt these processes, (2) exploration of the social mechanisms by which prosocial behavior is disseminated across a network, and (3) an indication of whether the alteration of contextual norms in favor of prosocial behavior can create a clustering process driven by prosocial behavior.

ELIGIBILITY:
Inclusion Criteria:

* All students in participating schools in the 7th grade (first year) and 8th grade (second year)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2064 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Substance use | twice a year for two years during 7th and 8th grades
  Tobacco, alcohol, and marijuana; actual use, intentions to use, willingness to use

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | twice a year for two years during 7th and 8th grades
  Externalizing, internalizing, and prosocial behavior
Engagement vs. Disaffection with Learning | twice a year for two years during 7th and 8th grades
  Behavioral and emotional engagement in learning
Classroom Life Scale | twice a year for two years during 7th and 8th grades
  Student academic support
University of Illinois Bully Scale | twice a year for two years during 7th and 8th grades
  Bullying and victimization

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Research Insititute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Van Ryzin MJ, Roseth CJ. Enlisting Peer Cooperation in the Service of Alcohol Use Prevention in Middle School. Child Dev. 2018 Nov;89(6):e459-e467. doi: 10.1111/cdev.12981. Epub 2017 Dec 19. PMID 29265358
- [Background] Van Ryzin MJ, Roseth CJ. Cooperative Learning in Middle School: A Means to Improve Peer Relations and Reduce Victimization, Bullying, and Related Outcomes. J Educ Psychol. 2018 Nov;110(8):1192-1201. doi: 10.1037/edu0000265. Epub 2018 Mar 1. PMID 30911200
- [Background] Van Ryzin MJ, Roseth CJ. Peer influence processes as mediators of effects of a middle school substance use prevention program. Addict Behav. 2018 Oct;85:180-185. doi: 10.1016/j.addbeh.2018.06.016. Epub 2018 Jun 13. PMID 29921538
- [Background] Van Ryzin MJ, Roseth CJ. Effects of cooperative learning on peer relations, empathy, and bullying in middle school. Aggress Behav. 2019 Nov;45(6):643-651. doi: 10.1002/ab.21858. Epub 2019 Aug 20. PMID 31432535
- [Derived] Lee DC, O'Brien KM, McCrabb S, Wolfenden L, Tzelepis F, Barnes C, Yoong S, Bartlem KM, Hodder RK. Strategies for enhancing the implementation of school-based policies or practices targeting diet, physical activity, obesity, tobacco or alcohol use. Cochrane Database Syst Rev. 2024 Dec 12;12(12):CD011677. doi: 10.1002/14651858.CD011677.pub4. PMID 39665378
- [Derived] Van Ryzin MJ, Roseth CJ. The Longitudinal Relationship Between Peer Relations and Empathy and their Joint Contribution to Reducing Bullying in Middle School: Findings from a Randomized Trial of Cooperative Learning. J Prev Health Promot. 2022 Apr;3(2):147-165. doi: 10.1177/26320770221094032. Epub 2022 May 5. PMID 36818659
- [Derived] Low S, Van Ryzin MJ, Roseth CJ. Peer learning can modify the reciprocal relationship between peer support and victimization in middle school. J Adolesc. 2023 Apr;95(3):524-536. doi: 10.1002/jad.12133. Epub 2022 Dec 22. PMID 36546511
- [Derived] Van Ryzin MJ, Cil G, Roseth CJ. Costs and benefits of cooperative learning as a universal school-based approach to adolescent substance use prevention. J Community Psychol. 2023 Jan;51(1):438-452. doi: 10.1002/jcop.22916. Epub 2022 Jul 8. PMID 35801306